CLINICAL TRIAL: NCT01120301
Title: NeuroThera® Efficacy and Safety Trial - 3 (NEST-3) A Double-blind, Randomized, Sham-controlled, Parallel Group, Multicenter, Pivotal Study to Assess the Safety and Efficacy of Transcranial Laser Therapy With the NeuroThera® Laser System for the Treatment of Acute Ischemic Stroke Within 24 Hours of Stroke Onset
Brief Title: Efficacy and Safety Trial of Transcranial Laser Therapy Within 24 Hours From Stroke Onset (NEST-3)
Acronym: NEST-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PhotoThera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTS-INT08-009
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2012-10

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Laser Therapy (Experimental)
  Interventions: Device: NeuroThera® Laser System
- Sham control procedure (Sham Comparator)
  Interventions: Device: NeuroThera® Laser System

INTERVENTIONS:
Device: NeuroThera® Laser System — Transcranial delivery of laser therapy or sham (no laser therapy) to the scalp

SUMMARY:
The purpose of this pivotal study is to demonstrate safety and efficacy of transcranial laser therapy (TLT) with the NeuroThera® Laser System in the treatment of subjects diagnosed with acute ischemic stroke. The initiation of the TLT procedure must be feasible for each subject between 4.5 and 24 hours of stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute ischemic stroke
2. Subject is not a candidate for treatment with neurothrombectomy
3. Initiation of the TLT procedure begins between 4.5 and 24 hours
4. Baseline NIHSS score range: 7-17
5. Full functional independence just prior to the present stroke episode
6. Negative pregnancy test in females of childbearing potential
7. Subject Informed Consent obtained prior to enrollment into this study

Exclusion Criteria:

1. Evidence of an intracranial, subdural, or subarachnoid hemorrhage
2. Acute ischemic strokes located exclusively in the brainstem, or cerebellum, or small deep infarctions, or massive hemispheric strokes
3. Seizure at stroke onset or within the 7 days prior to stroke onset
4. Sustained blood glucose >300 or <60 mg/dl
5. Sustained hypertension (SBP >220 mmHg or DBP >140 mmHg)
6. Sustained hypotension (SBP <80 mmHg or DBP <50 mmHg)
7. A presumed and/or confirmed septic embolus
8. History of CNS vascular disease (e.g. aneurysm, AVM) or history of CNS disease or damage (e.g. neoplasm or dementia) which may influence the subject's outcome assessment.
9. Head implant of any kind
10. Significant skin condition of the scalp (eg. psoriasis)
11. Use of any intravenous or intra-arterial thrombolytic medication
12. Use of any diagnostic or therapeutic interventional neurovascular procedure
13. Female who is pregnant or lactating or who is of childbearing potential and not using a medically acceptable method of birth control.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Disability assessed using the dichotomous modified Rankin Scale (mRS) | Day 90
Adverse event differences between transcranial laser therapy and sham | Day 90

SECONDARY OUTCOMES:
Distribution of scores across the ordinal mRS | Day 90
Binary outcome measure of the National Institute of Health Stroke Scale (bNIH) | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Werner Hacke, MD PhD, Study Chair — Heidelberg University; Justin Zivin, MD PhD, Study Chair — University of California, San Diego
Locations (60):
- United States (26):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Scripps Encinitas Hospital, Encinitas, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Stroke Center, Palo Alto, California
  - Munroe Regional Medical Center, Ocala, Florida
  - Gwinnett Medical Center, Duluth, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Parkview Hospital, Fort Wayne, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Minneapolis Clinic of Neurology, Robbinsdale, Minnesota
  - Saint Lukes Hospital, Kansas City, Missouri
  - University of Washington St. Louis, St Louis, Missouri
  - Mission Hospital/Mission Neurology Services, Asheville, North Carolina
  - University of North Carolina Healthcare, Chapel Hill, North Carolina
  - Guilford Neuro/The Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Erlanger Health System, Chattanooga, Tennessee
  - The Methodist Hospital, Houston, Texas
  - INOVA Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Harborview Medical Center, Seattle, Washington
- AKH Linz, Linz, Austria
- Canada (3):
  - University of Alberta Hospital - Walter C Mackenzie Health Science Center, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Trillium Health Centre, Mississauga, Ontario
- Helsinki University Central Hospital, Helsinki, Finland
- CHRU Lille-Hôpital Salengro, Lille, France
- Germany (18):
  - Neurologische Universitätsklinik Aachen, Aachen
  - Neurologische Klinik Bad Neustadt, Bad Neustadt an der Saale
  - Charité Campus Berlin Mitte (CCM), Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Heinrich-Heine-University of Düsseldorf, Düsseldorf
  - Neurologische Universitätsklinik Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Johann Wolfgang Goethe-University, Frankfurt am Main
  - Klinikum Frankfurt-Hochst, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinik und Poliklinik für Neurologie Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen
  - Johannes Wesling Klinikum Minden, Minden
  - Technische Universität München, München
  - Universitätsklinikum Münster, Münster
  - Kreisklinikum Siegen GmbH, Siegen
  - HSK, Dr. Horst Schmidt Klinik GmbH, Wiesbaden
- Hospital Nacional Dos de Mayo, Lima, Peru
- Spain (3):
  - Complejo Hospitalario Universitario Albacete, Albacete
  - University Hospital Vall D'Hebron, Barcelona
  - Hospital Universitari Dr Josep Trueta, Girona
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Sjukhuset i Lidköping, Lidköping
  - Kärnsjukhuset Skövde, Skövde
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Hacke W, Schellinger PD, Albers GW, Bornstein NM, Dahlof BL, Fulton R, Kasner SE, Shuaib A, Richieri SP, Dilly SG, Zivin J, Lees KR; NEST 3 Committees and Investigators. Transcranial laser therapy in acute stroke treatment: results of neurothera effectiveness and safety trial 3, a phase III clinical end point device trial. Stroke. 2014 Nov;45(11):3187-93. doi: 10.1161/STROKEAHA.114.005795. Epub 2014 Oct 7. PMID 25293665